CLINICAL TRIAL: NCT07019298
Title: Evaluation of the Success Rate of Endodontic Treatment Using Different Obturation Techniques and Root Canal Sealer Cements: A Randomized Controlled Trial
Brief Title: Success of Endodontic Treatment With Different Obturation Techniques and Sealer Cements
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Siena (Other)
Responsible Party: Principal Investigator, Simone Grandini, Prof, University of Siena
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HCCWC001
Record Dates: First submitted 2025-05-20; First posted 2025-06-13 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Pulpitis; Periapical Lesions; Periapical Periodontitis; Periapical Pathology
Keywords: Endodontics; Endodontic Sealer; Calcium Silicate-Based Sealer; Ah Plus
MeSH Terms: conditions — Pulpitis; Periapical Periodontitis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- AH Plus + Continuous Wave Condensation (Active Comparator): Root canal obturation using AH Plus (Dentsply Sirona, Charlotte, NC, USA) and the continuous wave technique with thermoplasticized gutta-percha
  Interventions: Procedure: AH Plus (Dentsply Sirona, Charlotte, NC, USA); Procedure: Continuous Wave Condensation
- AH Plus + Single Cone (Active Comparator): Root canal obturation using AH Plus and the single cone technique with cold gutta-percha.
  Interventions: Procedure: AH Plus (Dentsply Sirona, Charlotte, NC, USA); Procedure: Single Cone Technique
- NeoSealer Flo + Continuous Wave (Experimental): Root canal obturation using NeoSealer Flo (Avalon Biomed, Houston, TX, USA) and the continuous wave technique.
  Interventions: Procedure: NeoSealer Flo; Procedure: Continuous Wave Condensation
- NeoSealer Flo + Single Cone (Experimental): Root canal obturation using NeoSealer Flo and the single cone technique.
  Interventions: Procedure: NeoSealer Flo; Procedure: Single Cone Technique

INTERVENTIONS:
Procedure: AH Plus (Dentsply Sirona, Charlotte, NC, USA) — Root canal obturation using AH Plus (Dentsply Sirona, Charlotte, NC, USA), a resin-based sealer with low solubility and shrinkage. Used in combination with gutta-percha for root canal filling.
  Arms: AH Plus + Continuous Wave Condensation; AH Plus + Single Cone
Procedure: NeoSealer Flo — Root canal obturation using NeoSealer Flo (Avalon Biomed, Houston, TX, USA), a premixed bioceramic sealer based on calcium silicate. Used in combination with gutta-percha to enhance apical healing and biocompatibility.
  Arms: NeoSealer Flo + Continuous Wave; NeoSealer Flo + Single Cone
Procedure: Continuous Wave Condensation — A warm vertical compaction technique using heat-softened gutta-percha to obturate the canal in three dimensions. Considered the gold standard for achieving dense and homogenous root canal fillings.
  Arms: AH Plus + Continuous Wave Condensation; NeoSealer Flo + Continuous Wave
Procedure: Single Cone Technique — A cold hydraulic condensation technique using a single gutta-percha cone matched to the last rotary file, combined with a high-flow sealer. Designed for simplified obturation with minimal operator variability.
  Arms: AH Plus + Single Cone; NeoSealer Flo + Single Cone

SUMMARY:
The present study aims to compare the radiographic success of endodontic treatment using Orstavik's criteria between two sealers: AH Plus (Dentsply DeTrey, Konstanz, Germany) and Neosealer Flo (Avalon Biomed, Bradenton, Florida, USA), as well as between two obturation techniques: continuous wave and single cone. The study includes 270 patients, with a minimum follow-up period of 6 months. Clinical and radiographic variables will be assessed, including quality of obturation, lesion healing, and restoration. The study seeks to determine if the use of bioceramic sealer is effective regardless of the obturation technique used, highlighting the importance of clinical follow-up to evaluate endodontic treatment success.

ELIGIBILITY:
Inclusion Criteria:

Patients aged 18 years and older. Teeth with a diagnosis of pulpal necrosis or irreversible pulpitis. Informed consent provided for data usage.

Exclusion Criteria:

* Patients with systemic conditions that may impair healing (e.g., uncontrolled diabetes, immunosuppression).
* Teeth with root fractures, resorption, or open apices.
* Incomplete clinical or radiographic records.
* Cases with poor-quality radiographs or lack of standardization for evaluation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2029-06-01 (Estimated)

PRIMARY OUTCOMES:
Radiographic Success Based on Periapical Index (PAI) Criteria | Minimum 6 months after root canal treatment
  Radiographic outcome will be assessed using the Periapical Index (PAI) by Ørstavik et al. (1986), which categorizes periapical healing from 1 (normal periapical structures) to 5 (severe apical periodontitis).
  Success is defined as PAI scores of 1 or 2 (complete healing or healing in progress).
  Evaluations will be based on periapical radiographs (and CBCT when available) taken at follow-up after at least 6 months.
  The assessment will be performed by a calibrated blinded evaluator using reference radiographs.

SECONDARY OUTCOMES:
Clinical Success Based on Absence of Symptoms | Minimum 6 months after treatment
  Clinical success will be defined by the absence of pain, tenderness to percussion or palpation, swelling, mobility, and other signs of persistent infection.
  These parameters will be evaluated through standard clinical examination during follow-up visits.
Radiographic Success Based on CBCT Evaluation | Minimum 6 months after treatment
  When available, cone beam computed tomography (CBCT) images will be used to assess periapical healing.
  A modified periapical index (PAI-CBCT) will be used, evaluating the presence, size, and resolution of periapical radiolucencies.
  Lesion healing will be interpreted as success if there is full resolution or significant reduction in size compared to baseline.

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad Rey Juan Carlos, Madrid, Spain, Spain

IPD SHARING:
Plan to Share IPD: Undecided